CLINICAL TRIAL: NCT06081166
Title: A Study to Evaluate the Effect of Daily Doses of Obicetrapib Tablets on the Pharmacokinetics of Atorvastatin Calcium Tablets or Rosuvastatin Calcium Tablets in Healthy Adult Subjects
Brief Title: A Drug-drug Interaction Study Evaluating the PK Effects of Obicetrapib on Atorvastatin and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Collaborators: Pharma Medica Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TA-8995-11
Record Dates: First submitted 2023-10-03; First posted 2023-10-13 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Tablets; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Open-label, two-cohort, fixed sequence, drug-drug interaction study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- obicetrapib + atorvastatin (Active Comparator): Obicetrapib 10 mg tablets daily from Days 1-17 plus atorvastatin calcium 80 mg tablets on Day -4 and Day 12
  Interventions: Drug: Obicetrapib; Drug: Atorvastatin Calcium
- obicetrapib + rosuvastatin (Active Comparator): Obicetrapib 10 mg tablets daily from Days 1-17 plus rosuvastatin calcium 40 mg tablets on Day -4 and Day 12
  Interventions: Drug: Obicetrapib; Drug: Rosuvastatin Calcium

INTERVENTIONS:
Drug: Obicetrapib — obicetrapib 10 mg daily
  Other Names: tablets
Drug: Atorvastatin Calcium — Atorvastatin 80 mg
  Other Names: tablets
  Arms: obicetrapib + atorvastatin
Drug: Rosuvastatin Calcium — Rosuvastatin 40 mg
  Other Names: tablets
  Arms: obicetrapib + rosuvastatin

SUMMARY:
A study to evaluate impact of Obicetrapib on PK levels of Atorvastatin and Rosuvastatin

DETAILED DESCRIPTION:
A Study to Evaluate the Effect of Daily Doses of Obicetrapib Tablets on the Pharmacokinetics of Atorvastatin Calcium Tablets or Rosuvastatin Calcium Tablets in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Cohort 1 Healthy, non-smoking, male and female subjects, from 18 to 65 years of age Cohort 2 Healthy, non-smoking, male and female subjects of non-Asian origin, from 18 to 65 years of age
2. BMI ≥18.5 and ≤30 kg/m2
3. Females may be of childbearing or non-childbearing potential:

   * Childbearing potential:

     o Physically capable of becoming pregnant
   * Non-childbearing potential:

     * Surgically sterile (i.e., both ovaries removed, uterus removed, or bilateral tubal ligation); and/or
     * Postmenopausal (no menstrual period for at least 12 consecutive months without any other medical cause and FSH and LH values consistent with being postmenopausal).
4. Willing to use acceptable, effective methods of contraception.
5. Able to tolerate venipuncture.
6. Be informed of the nature of the study and give written consent prior to any study procedure

Exclusion Criteria:

1. Known history or presence of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Known or suspected carcinoma.
3. Known history or presence of hypersensitivity or idiosyncratic reaction to atorvastatin, rosuvastatin, obicetrapib, or any other drug substances with similar activity.
4. Known history or presence of chronic infectious disease, system disorders, organ dysfunction especially hypothyroidism, stroke or transient ischemic attack, myopathy, rhabdomyolysis, renal or hepatic disorders, diabetes, or obesity which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
5. Known history or presence of clinically significant lactose, galactose, or fructose intolerance.
6. Subjects of Asian origin (Cohort 2 only).
7. History of malabsorption within the last year or presence of clinically significant gastrointestinal (GI) disease.
8. Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.
9. History of drug or alcohol addiction requiring treatment.
10. Positive test result for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
11. Positive test result for urine drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, phencyclidine, and tricyclic antidepressants) or urine cotinine.
12. Difficulty consuming standard meals.
13. Use of tobacco or nicotine-containing products within 6 months prior to drug administration.
14. Females who:

    * Have used implanted, injected, intravaginal, or intrauterine hormonal contraceptives within 6 months prior to drug administration;
    * Have used oral or transdermal hormonal contraceptives within 21 days prior to drug administration;
    * Are pregnant (serum hCG consistent with pregnancy); or
    * Are breast-feeding.
15. Donation or loss of whole blood (including clinical trials):

    * ≥50 mL and <500 mL within 30 days prior to drug administration;
    * ≥500 mL within 56 days prior to drug administration.
16. Participation in a clinical trial that involved administration of an investigational medicinal product within 30 days prior to drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results.
17. On a special diet within 30 days prior to drug administration (e.g., liquid, protein, raw food diet).
18. Have had a tattoo or body piercing within 30 days prior to drug administration.
19. Have clinically significant findings in vital signs measurements.
20. Have clinically significant findings in a 12-lead ECG.
21. Have clinically significant abnormal laboratory values.
22. Have significant diseases.
23. Have clinically significant findings from a physical examination.
24. Use of any of the following within 30 days prior to drug administration:

    * Anticoagulants
    * Anti-fungals (e.g., voriconazole, itraconazole)
    * Anti-virals
    * Capmatinib
    * Cholestyramine
    * Colchicine
    * Cyclosporine
    * Darolutamide
    * Digoxin
    * Drugs known to induce/inhibit hepatic drug metabolism or alter GI pH/movement (e.g., omeprazole, ranitidine)
    * Fostamatinib
    * Inducers and inhibitors of CYP3A4
    * Inducers and inhibitors of breast cancer resistant protein
    * Inducers and inhibitors of OATP1B1/OATP1B3
    * Inducers and inhibitors of P-glycoprotein)
    * Macrolide antibiotic medications (e.g., erythromycin)
    * Niacin
    * Regorafenib
    * Statins
    * Tafamidis
    * Teriflunomide
    * Drugs that decrease levels of endogenous steroid hormones (e.g., ketoconazole, spironolactone, cimetidine)
    * Febuxostat
    * Fibrates (e.g., fenofibrate, gemfibrozil)
    * Warfarin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Measure atorvastatin/rosuvastatin levels in the blood | zero (0) to time of the last measurable analyte concentration (t), up to 22 days
  Measure atorvastatin/rosuvastatin concentrations via various analytical methods

CONTACTS AND LOCATIONS:
Overall Officials: Mark M Feldman, Principal Investigator — Pharma Medica Research, Inc.
Locations (1):
- Mark M Feldman, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kastelein JJP, Ditmarsch M, Hsieh A, Kling D, Walker A, Dicklin MR, Tayab Z, Bouhajib M, Davidson MH. A Drug-Drug Interaction Study Evaluating the Pharmacokinetic Consequences of Obicetrapib Therapy on Atorvastatin or Rosuvastatin Levels in Healthy Volunteers. Am J Cardiovasc Drugs. 2025 Sep;25(5):693-702. doi: 10.1007/s40256-025-00740-1. Epub 2025 Jun 26. PMID 40569335